CLINICAL TRIAL: NCT06119009
Title: New-onset Heart Blocks After Noncardiac Surgery: a Retrospective Study of More Than 280,000 Patients
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Hao Li, Director, Chinese PLA General Hospital
Other Study IDs: ChinesePLAGH301NBBB
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Heart Block; Risk Factor
Keywords: Postoperative new-onset heart blocks; Noncardiac surgery; Machine learning; Prediction model; Prognosis
MeSH Terms: conditions — Heart Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non- Heart blocks: The number of patients who did not suffered the heart blocks in the postoperative 1-year period
  Interventions: Other: non interventions
- Heart blocks: The number of patients who suffered the heart blocks in the postoperative 1-year period
  Interventions: Other: non interventions

INTERVENTIONS:
Other: non interventions

SUMMARY:
This study aimed to investigate new-onset heart blocks after noncardiac surgery, identify risk factors, and develop a prediction model.

DETAILED DESCRIPTION:
Objective: This study aimed to investigate new-onset heart blocks after noncardiac surgery, identify risk factors, and develop a prediction model.

Methods: A retrospective cohort study included 281,497 patients aged 18 or older who underwent noncardiac surgery at a single center between Jan 2008 and Aug 2019. The main outcome was postoperative new-onset heart blocks within one year, including atrioventricular and bundle blocks. Prognostic impact was assessed using Kaplan-Meier survival curves and time-dependent Cox regression analysis. Perioperative data was used for machine learning models (logistic regression, support vector machine, random forest, decision tree). Model performance was measured using the area under the receiver operating characteristic curve (AUC).

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 yrs undergoing noncardiac surgery at the First Medical Center of the Chinese People's Liberation Army General Hospital (PLAGH) from January 1, 2008 to August 1, 2019.

Exclusion Criteria:

* surgical duration of less than 30 minutes
* incomplete data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data were gathered from electronic medical records (EMRs) for all patients undergoing noncardiac surgery at the First Medical Center of the Chinese People's Liberation Army General Hospital (PLAGH) from January 1, 2008 to August 1, 2019. Patients with a surgical duration of less than 30 minutes or age <18 years were excluded. Input data elements were extracted from the patient anesthesia and medical records. The survival data one year after surgery were obtained from medical records and telephone follow-up records confirmed by the Chinese Center for Disease Control and Prevention (CCDC)
Sampling Method: Non-Probability Sample
Enrollment: 281497 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
New-onset heart blocks | within one year after surgery
  The number of new-onset heart blocks within one year after surgery, including first-, second-, and third-degree AV blocks and left- and right-branch bundle blocks